CLINICAL TRIAL: NCT01218945
Title: Development of Bone Grafts Using Adipose Derived Stem Cells and Different Scaffolds: Impact of Pre-engineered Capillaries in Critical Size Grafts
Brief Title: Development of Bone Grafts Using Adipose Derived Stem Cells and Different Scaffolds
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: Bone-ZH09
Record Dates: First submitted 2010-09-29; First posted 2010-10-11 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight | interventions — Cell Culture Techniques

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human adipose-derived stem cells from human fat
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fat Removal: Patients undergoing surgical fat removal
  Interventions: Procedure: Cell Culture

INTERVENTIONS:
Procedure: Cell Culture — Aim of this study is to isolate and cultivate fat-derived progenitor cells and differentiation into osteoblasts. Therefore, our research idea is to pre-engineer large synthetic bone grafts and study the vascularization process in vivo.

SUMMARY:
The repair of large osseous defects remains still unsolved. Aim of this study is to isolate and cultivate fat-derived progenitor cells and differentiation into osteoblasts. Therefore, our research idea is to pre-engineer large synthetic bone grafts and study the vascularization process in vivo.

ELIGIBILITY:
Inclusion criteria:

* German-speaking patients aged 18-70 admitted to the Clinic of Reconstructive surgery for reconstructive surgery and fat-excision.

Exclusion criteria:

* Drug-abuse, neoplasia and metabolic disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted for reconstructive surgery
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Calcagni, MD, Principal Investigator — University Hospital Zurich, Clinic of Reconstructive Surgery
Locations (1):
- University Hospital Zurich, Clinic of Reconstructive Surgery, Zurich, Canton of Zurich, Switzerland